CLINICAL TRIAL: NCT02857790
Title: MRI Before and After Coronary Angioplasty With Rotational Atherectomy
Brief Title: Glasgow MRI and Rotablation Study
Acronym: GlaMoRouS
Status: Completed | Type: Observational
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: University of Glasgow (Other); Cardiovascular Research Foundation, New York (Other); Medical Research Scotland (Unknown); Chief Scientist Office of the Scottish Government (Other Government); Scottish Funding Council (Unknown); Engineering and Physical Sciences Research Council (EPSRC) (Unknown)
Responsible Party: Principal Investigator, Margaret McEntegart, Consultant Cardiologist, NHS National Waiting Times Centre Board
Other Study IDs: 11/CARD/18
Record Dates: First submitted 2016-07-20; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
Keywords: Rotablation; High speed rotational atherectomy; Type IV myocardial infarction; Cardiac magnetic resonance imaging; CMR; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Percutaneous coronary intervention (PCI) with adjunctive high speed rotational atherectomy (HSRA) is commonly used to treat complex and calcified coronary artery stenoses. Theoretically, HSRA may have deleterious effects on the coronary microcirculation and result in peri-procedural myocardial infarction (Type 4a MI).

This study is assessing the effects of HSRA PCI using serial multi-parametric stress perfusion cardiac magnetic resonance imaging (CMR) (1.5 Tesla MAGNETOM Avanto, Siemens Healthcare). The study will prospectively enrol up to 75 patients (minimum completed cohort of 50 patients) undergoing elective HSRA PCI and performing multi-parametric CMR at 3 time-points: before HSRA, 1 week post-HSRA, and 6 months post-HSRA. Myocardial perfusion will be assessed using pharmacological stress with intravenous adenosine (140 micrograms/kg/min) at each time point. High-sensitivity cardiac troponin (hsTn) and ECGs will be performed post-HSRA.

DETAILED DESCRIPTION:
High Speed Rotational atherectomy (HSRA) is a technique used during angioplasty in the treatment of calcified coronary arteries. Rotablation debulks resistant calcium in the coronary artery plaque thus facilitating stent deployment and expansion. The atherectomy technique involves a rotating diamond-tipped burr which breaks down the calcium into small particles which are washed forward by the blood flow into the smaller coronary branches supplying the heart muscle. The dispersed calcium particles may block these smaller blood vessels, interrupting blood flow to an extent that may result in heart muscle damage. When this injury becomes detectable clinically, with symptoms, ECG changes and increased troponin, an iatrogenic type IV myocardial infarction (MI) is diagnosed.

Cardiac magnetic resonance imaging (CMR) is the gold standard method for imaging the heart providing detailed information on cardiac function and muscle injury.

This is a prospective cohort observational study of 60 patients undergoing coronary angioplasty with rotational atherectomy.

The aim of the study is to investigate myocardial injury revealed by paired CMR scans before and after rotational atherectomy.

The hypothesis is that following rotational atherectomy, displacement of calcified particles cause microvascular obstruction leading to reduced perfusion. Since myocardial perfusion and pump function are linked, as myocardial perfusion is reduced after atherectomy, so myocardial contractility (i.e. strain) will reduce. In a second analysis, computer modelling will be used to integrate the different types of CMR information to better understand the spatial, temporal and pathological evolution of myocardial infarction (www.softmech.org). The further hypothesis is that despite CMR detectable infarction the incidence of clinical type IV MI will be low.

CMR scans will be performed 1 week before, 1 week and 6 months post rotablation. Cardiac troponin and ECGs will be performed post rotablation to determine the incidence of type IV MI.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina
* Indication for PCI with rotablation

Exclusion Criteria:

* Other major systemic illness
* Contra-indication to CMR
* Pregnancy
* CKD (eGFR<30)
* Pre-existing infarct in culprit vessel territory on ECG, echo or baseline CMR
* Chronic total occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Near consecutive eligible patients undergoing elective PCI with rotablation.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2012-03; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in circumferential myocardial strain | 1 week and 6 months post-rotablation

SECONDARY OUTCOMES:
Incidence of CMR detected de novo late gadolinium enhancement | 1 week and 6 months post-rotablation
Incidence of type IV myocardial infarction | 6-12 hours post-rotablation
Change in ischaemic burden | 1 week and 6 months post-rotablation
Change in left ventricular ejection fraction (LVEF) | 1 week and 6 months post-rotablation
Change in left ventricular (LV) volumes | 1 week and 6 months post-rotablation
Index of Microcirculatory Resistance (IMR) | Intra-procedural baseline, intra-procedural post-rotablation, and intra-procedural post-stenting
Minimum Stent Area (MSA) | Intra-procedural post-rotablation

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McEntegart, Principal Investigator — Golden Jubilee National Hospital; Colin Berry, Principal Investigator — University of Glasgow

IPD SHARING:
Plan to Share IPD: No